CLINICAL TRIAL: NCT01210716
Title: Evaluation of Therapeutic Plasma Exchange (TPE) Procedure Using the AMICUS Device
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fenwal, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: FCRP- 0210
Record Dates: First submitted 2010-09-26; First posted 2010-09-28 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Autoimmune Diseases; Renal Disorders; Hematologic Disorders; Oncologic Disorders
Keywords: Therapeutic plasma exchange; Autoimmune diseases; Kidney transplant; Hematologic disorders; Monoclonal gammopathy; Neurologic disorders
MeSH Terms: conditions — Autoimmune Diseases; Kidney Diseases; Hematologic Diseases; Paraproteinemias; Nervous System Diseases | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMICUS Therapeutic plasma exchange, TPE (Experimental): Patients are randomized to either TPE on AMICUS or Spectra.
  Interventions: Device: Therapeutic plasma exchange
- Spectra Therapeutic plasma exchange, TPE (Active Comparator): Patients are randomized to either TPE on AMICUS or Spectra.
  Interventions: Device: Therapeutic plasma exchange

INTERVENTIONS:
Device: Therapeutic plasma exchange — Patients are randomized to either Therapeutic plasma exchange procedures on AMICUS or Spectra first. The second procedure (based on time interval determined by physician) will be completed on the other instrument.
  Other Names: TPE

SUMMARY:
This study will evaluate the use of the AMICUS device in patients where Therapeutic Plasma Exchange (TPE) is prescribed by their physicians.

DETAILED DESCRIPTION:
Therapeutic plasma exchange (TPE) is intended for efficient removal of circulating plasma, with the return of replacement fluids to the patient. In the majority of cases, the treatment goal is to selectively remove the substance directly responsible for the patient's disease process.

Fenwal's AMICUS separator platform is a centrifuge-based apheresis system which collects the blood components of interest and returns the remaining blood components along with saline back to a donor/patient. The device has been cleared for the following:

* The collection of platelets and plasma in Japan, Europe and the US (BK960005), 1996.
* The collection of mononuclear cells (MNCs) in the US (BK000047), 2002.
* The collection of a concurrent red blood cell (cRBC) product collected in ACD-A anticoagulant and stored in ADSOL® Preservation Solution (BK000039), 2002.

Fenwal has developed a new protocol on the AMICUS separator that enables the device to perform TPE procedures. The procedure is similar to the FDA cleared platelet and concurrent plasma collections, except that in TPE procedures the majority of plasma is retained and the red blood cells (RBCs), white blood cells (WBC) and the majority of the platelets are returned to the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Medically stable patients undergoing more than one TPE procedure who have provided signed informed consent prior to participation.
2. A physician's prescription for TPE for various non-emergent conditions.
3. Test and Control TPE procedures that would be expected to be completed within approximately five weeks.

Exclusion Criteria:

1. Patients under 18 years old.
2. Patients on an ACE inhibitor medication should discontinue use of this medication in accordance with institutional practices.
3. Patients with altered mental status that would prohibit the giving and understanding of informed consent.
4. Patients who have experienced a serious adverse event associated with the first TPE clinical study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peyton Metzel, PhD, Study Chair — Fenwal, Inc.
Locations (4):
- United States (4):
  - Yale University School of Medicine, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota
  - University of Virginia, Charlottesville, Virginia
  - BloodCenter of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened enrollment on Sept 2010 at three hospitals-Yale New Haven Hospital, Mayo Clinic and University of Virginia Health System. A 4th site, BloodCenter of Wisconsin opened enrollment April,2011.
Pre-assignment Details: Patients were required to complete two (2) procedures. First procedure was randomized to either Therapeutic plasma exchange on active comparator (AMICUS) or current device (Spectra). The second procedure was completed within approximately 5 weeks on the other device per physician prescription.
Groups:
- Spectra First, Then AMICUS: Patients randomized to Control (Spectra) procedure first. Second procedure performed was Test (AMICUS).
- AMICUS First, Then Spectra: Patients randomized to Test (AMICUS) procedure first. Second procedure performed was Control (Spectra).
Period: First TPE Procedure
Arm/Group | Spectra First, Then AMICUS | AMICUS First, Then Spectra
Started | 20 | 17
Completed | 18 | 15
Not Completed | 2 | 2
Period: Second TPE Procedure
Arm/Group | Spectra First, Then AMICUS | AMICUS First, Then Spectra
Started | 18 | 15
Completed | 15 | 15
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Demographics were reported for the evaluable patient population.
Groups:
- Overall Study Population: Includes groups randomized to receive Spectra first and AMICUS first.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 50.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Percent Efficiency of Plasma Removal During the Therapeutic Plasma Exchange Procedure
Description: The calculation is based on the volume of plasma that was processed through the machine compared to the volume of patient plasma that was actually removed during the procedure.
  Plasma Efficiency = (plasma removed/plasma processed)*100
Time Frame: After completion of the TPE procedure.
Population: A total of 37 patients who consented and enrolled started the 1st procedure. Of these 37 patients, 33 patients completed the 1st procedure and started a 2nd procedure. Three patients did not complete the second procedure resulting in 30 patients with completed paired Test and Control procedures.
Measure: Mean (Full Range); unit: percentage of plasma removal efficiency
Groups:
- AMICUS (Test): Each evaluable patient underwent one complete TPE procedure on the AMICUS separator.
- Spectra (Control): Each evaluable patient underwent one complete TPE procedure on the COBE Spectra separator.
Arm/Group | AMICUS (Test) | Spectra (Control)
Number analyzed (Participants) | 30 | 30
percentage of plasma removal efficiency | 81.9 [68 to 96] | 75.2 [61 to 88]
Statistical Analysis 1: Comparison: AMICUS (Test) vs Spectra (Control); A one-sample t-test on the mean of paired differences was used to evaluate the primary objective. Sample size was determined using historical data and the 95% chi-square upper confidence limit on the observed standard deviation of the paired differences. A minimum sample of 27 pairs was required to demonstrate the AMICUS procedure to be non-inferior to Spectra with a mean efficiency of plasma removal with a non-inferiority margin of 15% with at least 97.5% (one-sided) confidence and 90% power; Test type: Non-Inferiority or Equivalence — If the lower 97.5% confidence limit on the mean of the paired differences is greater than -15% of the Control group mean (i.e., p-value <=0.05), then the Test group will be considered non-inferior in the primary efficacy parameter to Control at the margin of 15%; p < 0.001, paired t-test; Mean Difference (Final Values) = 6.69, 95% CI 1-sided [lower limit 4.0], Standard Deviation 6.970

2. Secondary Outcome: Safety Measured by Adverse Events During the TPE Procedure
Time Frame: Adverse events were collected during each TPE procedure.
Population: Adverse events were summarized for enrolled subjects per protocol. 7 out of 37 enrolled subjects experienced adverse events during the study with a total of 12 adverse events reported.
Measure: Number; unit: participants
Arm/Group | Overall Study Population
Number analyzed (Participants) | 37
participants | 7 [61 to 88]

ADVERSE EVENTS:
Arm/Group | Overall Study Population
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 7/37
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study Population (N=37)
Dizzy/Light-Headed (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Infiltration (Skin and subcutaneous tissue disorders) | 1 (1)
Chills (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Rigors (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of data and/or information derived from the study requires prior review and approval by Sponsor.